CLINICAL TRIAL: NCT02490527
Title: Effects of Epicatechin on Patients With Statin-induced Mitochondrial Dysfunction and Impaired Exercise Capacity
Brief Title: Effects of Epicatechin on Statins for Mitochondrial Dysfunction and Impaired Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCSD IRB 150171
Record Dates: First submitted 2015-06-17; First posted 2015-07-07 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Statin Intolerance
Keywords: myopathy; muscular weakness; cramping; fatigue
MeSH Terms: conditions — Muscular Diseases; Muscle Weakness; Spasm; Fatigue | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin only (Placebo Comparator): The subject will consume simvastatin (40mg) and placebo once daily for 3 months.
  Interventions: Drug: Simvastatin (40mg); Other: Placebo
- Statin and epicatechin (Experimental): The subject will consume simvastatin (40mg) and pure epicatechin capsules (50mg) once daily for 3 months.
  Interventions: Dietary Supplement: Pure epicatechin capsules (50mg); Drug: Simvastatin (40mg)

INTERVENTIONS:
Dietary Supplement: Pure epicatechin capsules (50mg) — Epicatechin is a compound found naturally in dark chocolate.
  Arms: Statin and epicatechin
Drug: Simvastatin (40mg) — A cholesterol-lowering medication that blocks the production of cholesterol.
Other: Placebo — A substance that has no therapeutic effect and will act as a control.
  Arms: Statin only

SUMMARY:
The purpose of this study is to gain insight into the side-effects of statin consumption, and assess the ability of epicatechin (a compound in dark chocolate) to counteract or reverse these changes. The investigators' prior research has shown that epicatechin can improve skeletal muscle structure and mitochondrial (which gives us energy) structure.

DETAILED DESCRIPTION:
Patient Inclusion Criteria:

1. Must be between 30-75 years of age.
2. Must have a VO2max greater than 18 ml/kg/min(non-sedentary individuals).
3. Subjects with LDL>100mg/dL (or on drug treatment)
4. Subjects without a prior cerebrovascular event (example: stroke)
5. Subjects without a prior cardiovascular event (example: heart attack)

Patient Exclusion Criteria:

1. Liver, thyroid, or kidney disease.
2. Currently taking drugs that interfere with statin metabolism (calcium channel blockers, colchicine etc.).
3. Acute or chronic infectious disease; autoimmune/inflammatory disease, cancer, COPD, anemia, diabetes, psychiatric illness.
4. Non-smokers, prior smokers, or illicit drug users with abstinence >1 year.
5. Subjects taking blood thinners (Coumadin, xarelto, pradaxa, Plavix, effient, apixiban, etc) will be excluded. If subjects are taking aspirin for routine prevention they will be asked to hold aspirin for 7 days prior to biopsy. Routine prevention means that the patients are taking aspirin to reduce their risks, but do not have established cardiovascular disease.
6. History of previous knee surgery and active history of knee pain or neuromuscular disease are exclusions as they are known to affect muscle structure and function.

The study will be a double blind placebo controlled study where subjects will be randomized to either of two groups:

1. Simvastatin 40 mg + placebo once daily (statin only group) for 3 months
2. Simvastatin 40 mg + Epi 50 mg once daily (statin + Epi group) for 3 months

ELIGIBILITY:
Patient Inclusion Criteria:

* Must be between 30-75 years of age
* LDL>100mg/dL (or on drug treatment)
* VO2 max greater than 25 ml/kg/min

Patient Exclusion Criteria:

* Liver or kidney disease
* Currently taking drugs that interfere with statin metabolism
* Currently taking blood thinners
* Acute or chronic infectious disease; autoimmune/inflammatory disease, cancer, COPD, anemia, psychiatric illness, insulin-dependent diabetes
* smokers or illicit drug users
* adverse cardiovascular event (ex: heart attack)
* history of knee surgery or active history of knee pain

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in Functional Capacity | Baseline and 3 months
  Cardiopulmonary exercise protocol will be used to measure VO2max to assess functional capacity.

OTHER OUTCOMES:
Changes in Blood-Based Biomarkers | Baseline and 3 months
  Biomarker levels in the blood will be evaluated for correlation with changes in the skeletal muscle mitochondrial structure and function.
Composite Outcome: Changes in Skeletal Muscle Structure and Protein Levels | Baseline and 3 months
  The optional skeletal muscle biopsies will be examined by electron microscopy to determine change in skeletal muscle structure. Western blots will be done to look for changes in protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Taub PR, Ramirez-Sanchez I, Ciaraldi TP, Perkins G, Murphy AN, Naviaux R, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. Alterations in skeletal muscle indicators of mitochondrial structure and biogenesis in patients with type 2 diabetes and heart failure: effects of epicatechin rich cocoa. Clin Transl Sci. 2012 Feb;5(1):43-7. doi: 10.1111/j.1752-8062.2011.00357.x. Epub 2011 Nov 7. PMID 22376256
- [Background] Yamazaki KG, Taub PR, Barraza-Hidalgo M, Rivas MM, Zambon AC, Ceballos G, Villarreal FJ. Effects of (-)-epicatechin on myocardial infarct size and left ventricular remodeling after permanent coronary occlusion. J Am Coll Cardiol. 2010 Jun 22;55(25):2869-76. doi: 10.1016/j.jacc.2010.01.055. PMID 20579545
- [Background] Nogueira L, Ramirez-Sanchez I, Perkins GA, Murphy A, Taub PR, Ceballos G, Villarreal FJ, Hogan MC, Malek MH. (-)-Epicatechin enhances fatigue resistance and oxidative capacity in mouse muscle. J Physiol. 2011 Sep 15;589(Pt 18):4615-31. doi: 10.1113/jphysiol.2011.209924. Epub 2011 Jul 25. PMID 21788351
- [Background] Ramirez-Sanchez I, Nogueira L, Moreno A, Murphy A, Taub P, Perkins G, Ceballos GM, Hogan M, Malek M, Villarreal F. Stimulatory effects of the flavanol (-)-epicatechin on cardiac angiogenesis: additive effects with exercise. J Cardiovasc Pharmacol. 2012 Nov;60(5):429-38. doi: 10.1097/FJC.0b013e318269ae0d. PMID 22833114
- [Background] Ramirez-Sanchez I, Taub PR, Ciaraldi TP, Nogueira L, Coe T, Perkins G, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. (-)-Epicatechin rich cocoa mediated modulation of oxidative stress regulators in skeletal muscle of heart failure and type 2 diabetes patients. Int J Cardiol. 2013 Oct 9;168(4):3982-3990. doi: 10.1016/j.ijcard.2013.06.089. Epub 2013 Jul 17. PMID 23870648
- [Background] Taub PR, Ramirez-Sanchez I, Ciaraldi TP, Gonzalez-Basurto S, Coral-Vazquez R, Perkins G, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. Perturbations in skeletal muscle sarcomere structure in patients with heart failure and type 2 diabetes: restorative effects of (-)-epicatechin-rich cocoa. Clin Sci (Lond). 2013 Oct;125(8):383-9. doi: 10.1042/CS20130023. PMID 23642227
- [Background] Barnett CF, Moreno-Ulloa A, Shiva S, Ramirez-Sanchez I, Taub PR, Su Y, Ceballos G, Dugar S, Schreiner G, Villarreal F. Pharmacokinetic, partial pharmacodynamic and initial safety analysis of (-)-epicatechin in healthy volunteers. Food Funct. 2015 Mar;6(3):824-33. doi: 10.1039/c4fo00596a. PMID 25598082
- [Background] Ortiz-Vilchis P, Yamazaki KG, Rubio-Gayosso I, Ramirez-Sanchez I, Calzada C, Romero-Perez D, Ortiz A, Meaney E, Taub P, Villarreal F, Ceballos G. Co-administration of the flavanol (-)-epicatechin with doxycycline synergistically reduces infarct size in a model of ischemia reperfusion injury by inhibition of mitochondrial swelling. Eur J Pharmacol. 2014 Dec 5;744:76-82. doi: 10.1016/j.ejphar.2014.09.042. Epub 2014 Oct 2. PMID 25281837
- [Background] Gutierrez-Salmean G, Ciaraldi TP, Nogueira L, Barboza J, Taub PR, Hogan MC, Henry RR, Meaney E, Villarreal F, Ceballos G, Ramirez-Sanchez I. Effects of (-)-epicatechin on molecular modulators of skeletal muscle growth and differentiation. J Nutr Biochem. 2014 Jan;25(1):91-4. doi: 10.1016/j.jnutbio.2013.09.007. Epub 2013 Oct 18. PMID 24314870
- [Derived] Ormiston CK, Pazargadi A, Rosander A, Ceballos G, Villarreal F, Taub PR. Enhancement of Statin Effects on Lipid Lowering and Reduction of Cardiovascular Risk Score by (-)-Epicatechin in Proof-of-Concept Pilot Study. Clin Transl Sci. 2025 May;18(5):e70236. doi: 10.1111/cts.70236. PMID 40387782